CLINICAL TRIAL: NCT06232382
Title: A Comparison of Hypnosis and Mindfulness on Reducing Pain in Chronic Pain Patients: A Randomized Controlled Study
Brief Title: A Comparison of Hypnosis and Mindfulness on Reducing Pain in Chronic Pain Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Sarocha Watatham, Co-investigator, Pain Fellow, Siriraj Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Si 912/2023
Record Dates: First submitted 2023-12-30; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Hypnosis, Mindfulness Meditation

STUDY DESIGN:
Intervention Model Description: 1. Audio hypnosis (HYP)
  2. Audio mindfulness (MM)
  3. A control condition (a voice reading neutral text)
Who Masked: Investigator, Outcomes Assessor
Masking Description: * Participants will be blind to the study hypotheses.
  * To keep the experimenter blind, the participants will not reveal what they hear in the audios.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hypnosis Audio (Experimental): 20 minutes audio
  Interventions: Other: Hypnosis audio
- Mindfulness meditation (Experimental): 20 minutes audio
  Interventions: Other: Mindfulness meditation audio
- Natural text audio (Placebo Comparator): 20 minutes audio
  Interventions: Other: Natural text audio (control audio)

INTERVENTIONS:
Other: Hypnosis audio — * After informed consent was obtained and baseline assessment, patients will be randomly assigned to one of the three conditions in 20 minutes:
    1. Audio hypnosis (HYP)
    2. Audio mindfulness (MM)
    3. A control condition (a voice reading neutral text) These audios will be produced together with hypnotherapist in Thailand, psychiatrist and researchers.
  * The randomization process will be performed using a computerized random sequence generator.
  * The patient listens to "Hypnosis" audio recording through headphones in a private room.
  * Participants will be blind to the study hypotheses.
  * To keep the experimenter blind, the participants will not reveal what they hear in the audios.
  * Pain intensity will be assessed both at pre- and post-session (5 minutes).
  * Secondary outcomes will be assessed at pre- and post-session by the questionnaires (5 minutes).
  * Post-session quality of sleep will be assessed by telephone interview 1 day after session.
  Arms: Hypnosis Audio
Other: Mindfulness meditation audio — * After informed consent was obtained and baseline assessment, patients will be randomly assigned to one of the three conditions in 20 minutes:
    1. Audio hypnosis (HYP)
    2. Audio mindfulness (MM)
    3. A control condition (a voice reading neutral text) These audios will be produced together with hypnotherapist in Thailand, psychiatrist and researchers.
  * The randomization process will be performed using a computerized random sequence generator.
  * The patient listens to "Mindfulness Meditation" audio recording through headphones in a private room.
  * Participants will be blind to the study hypotheses.
  * To keep the experimenter blind, the participants will not reveal what they hear in the audios.
  * Pain intensity will be assessed both at pre- and post-session. (5 minutes)
  * Secondary outcomes will be assessed at pre- and post-session by the questionnaires. (5 minutes)
  * Post-session quality of sleep will be assessed by telephone interview 1 day after session.
  Arms: Mindfulness meditation
Other: Natural text audio (control audio) — * After informed consent was obtained and baseline assessment, patients will be randomly assigned to one of the three conditions in 20 minutes:
    1. Audio hypnosis (HYP)
    2. Audio mindfulness (MM)
    3. A control condition (a voice reading neutral text) These audios will be produced together with hypnotherapist in Thailand, psychiatrist and researchers.
  * The randomization process will be performed using a computerized random sequence generator.
  * The patient listens to "Control" audio recording through headphones in a private room.
  * Participants will be blind to the study hypotheses.
  * To keep the experimenter blind, the participants will not reveal what they hear in the audios.
  * Pain intensity will be assessed both at pre- and post-session. (5 minutes)
  * Secondary outcomes will be assessed at pre- and post-session by the questionnaires. (5 minutes)
  * Post-session quality of sleep will be assessed by telephone interview 1 day after session.
  Arms: Natural text audio

SUMMARY:
The goal of this randomized controlled study is to evaluate the efficacy of an audio session of hypnosis and mindfulness meditation for providing immediate pain relief in individuals with chronic pain from Thailand. The main question[s] it aims to answer are:

• What effects do hypnosis and mindfulness meditation on reducing pain in chronic pain patients? Participants will

* Be randomly assigned to one of the three conditions in 20 minutes: Audio hypnosis, Audio mindfulness, A control condition
* Be blind to the study hypotheses.
* To keep the experimenter blind, the participants will not reveal what they hear in the audio.
* Pain intensity will be assessed both at pre- and post-session.
* Secondary outcomes will be assessed at pre- and post-session by the questionnaires.
* Post-session quality of sleep will be assessed by telephone interview 1 day after the session.

Primary outcome: Current pain intensity (using a 0 - 10 numerical rating scale) Secondary outcome

* Anxiety at pre and post-session using a 0-10 numerical rating scale
* 0-10 numerical rating scale assessing average, worst, and least pain intensity experienced during the sessions
* 1-5 categorical scale of treatment satisfaction assessed at post-treatment
* Quality of sleep using the Thai version of the Patient-Reported Outcomes Measurement Information System-29 (T-PROMIS-29) sleep disturbance section (4 items) at pre-session and 1 day after a session (by telephone interview)
* Duration of benefit The proposed measures of these variables have all been used successfully in prior clinical trials in samples of individuals with pain from Thailand.

ELIGIBILITY:
Inclusion Criteria:

1. Being ≥ 18 years old
2. Having chronic, non cancer pain (i.e., reporting bothersome pain for at least 50% of the days during the last three months)
3. Nociceptive, neuropathic, nociplastic pain characteristic
4. Endorsing having current pain intensity of ≥ 4 on a 0 to 10 Numerical Rating Scale
5. Being able to read, speak, and understand Thai

Exclusion Criteria:

1. Having significant hearing loss that would interfere with being able to hear the study audio
2. Having significant cognitive dysfunction, physical disability, or severe mood disturbance (e.g., significant anger or high lability) that would interfere with being able to participate in the study procedures
3. Cancer-related pain or cancer patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity | Baseline (immediately prior to intervention), 5 minutes after the intervention
  Current pain intensity will be assessed using a 0 - 10 numerical rating scale with 0 = "No pain" and 10 = "Pain as bad as it could be."

SECONDARY OUTCOMES:
Change in anxiety | Baseline (immediately prior to intervention), 5 minutes after the intervention
  Anxiety at pre- and post-session using a 0-10 numerical rating scale with 0 = "No anxiety" and 10 = "Anxiety as bad as it could be."
Average, worst, and least pain intensity experienced during the sessions | 5 minutes after the intervention
  0-10 numerical rating scale with 0 = "No pain" and 10 = "Pain as bad as it could be." assessing average, worst, and least pain intensity experienced during the sessions
Satisfaction | 5 minutes after intervention
  1-5 categorical scale of treatment satisfaction assessed at post-treatment
  - "Not at all Satisfied," "Partly Satisfied," "Satisfied," "More than Satisfied," "Very Satisfied," numbering 1 to 5 as an interval scale.
Change in quality of sleep | Baseline (immediately prior to intervention) and 24 hours after session (by telephone interview)
  Quality of sleep using the Thai version of the Patient-Reported Outcomes Measurement Information System-29 (T-PROMIS-29) sleep disturbance section (4 items)
  - Minimum score = 4, Maximum score = 20 (higher scores mean a worse outcome)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adachi T, Fujino H, Nakae A, Mashimo T, Sasaki J. A meta-analysis of hypnosis for chronic pain problems: a comparison between hypnosis, standard care, and other psychological interventions. Int J Clin Exp Hypn. 2014;62(1):1-28. doi: 10.1080/00207144.2013.841471. PMID 24256477
- [Background] Hilton L, Hempel S, Ewing BA, Apaydin E, Xenakis L, Newberry S, Colaiaco B, Maher AR, Shanman RM, Sorbero ME, Maglione MA. Mindfulness Meditation for Chronic Pain: Systematic Review and Meta-analysis. Ann Behav Med. 2017 Apr;51(2):199-213. doi: 10.1007/s12160-016-9844-2. PMID 27658913
- [Background] Thuma K, Ditsataporncharoen T, Arunpongpaisal S, Siripul P. Hypnosis as an Adjunct for Managing Pain in Head and Neck Cancer Patients Post Radiotherapy. J Med Assoc Thai. 2016 Aug;99 Suppl 5:S141-7. PMID 29906024
- [Background] Jensen MP, Sherlin LH, Askew RL, Fregni F, Witkop G, Gianas A, Howe JD, Hakimian S. Effects of non-pharmacological pain treatments on brain states. Clin Neurophysiol. 2013 Oct;124(10):2016-24. doi: 10.1016/j.clinph.2013.04.009. Epub 2013 May 22. PMID 23706958
- [Result] Cimmino MA, Ferrone C, Cutolo M. Epidemiology of chronic musculoskeletal pain. Best Pract Res Clin Rheumatol. 2011 Apr;25(2):173-83. doi: 10.1016/j.berh.2010.01.012. PMID 22094194